CLINICAL TRIAL: NCT06179420
Title: The Effectiveness of Advanced Decision Support Tool (OPT-IVF) for IVF Treatment
Status: Not yet recruiting | Type: Observational
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Azrai Abu, Associate Prof, National University of Malaysia
Other Study IDs: UKMPPI/111/8/JEP-2023-735
Record Dates: First submitted 2023-12-10; First posted 2023-12-21 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Fertility Issues
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- standard IVF regime protocol based on clinician decision: The dosage of gonadotrophin and time of transvaginal ultrasound decided by clinician
  Interventions: Other: total cumulative gonadotrophin usage
- clinical decision support tool, Opt-IVF for IVF regime protocol: The dosage of gonadotrophin and time of transvaginal ultrasound decided by a clinical decision support tool ( OPt -IVF)
  Interventions: Other: total cumulative gonadotrophin usage

INTERVENTIONS:
Other: total cumulative gonadotrophin usage — total dosage in IU
  Other Names: number of matured oocytes; number of qood quality blastocyst

SUMMARY:
This prospective study is subject to approval of institutional medical research ethics committee. Patient undergoing second cycle IVF will be enrolled into the intervention group. Intervention involved using a clinical decision support tool, Opt-IVF to guide gonadotrophins dosing and trigger dates for a personalized controlled ovarian stimulation cycle based on the distribution of follicle sizes on day 1 and day 5, and hormone dosages given on day 1 to 4.

Patients will undergo transvaginal ultrasound exam on day 1 and day 5 of the cycle to determine the number and size of follicles present. The data is used in the Opt-IVF decision support tool to suggest Gonadotropin dosage for D5 and beyond and to recommend the antagonist start day and trigger day.

Clinical investigators will not override the Opt-IVF recommended dosage in any patients.

DETAILED DESCRIPTION:
The total dosage of gonadotrophin, number of good quality oocytes and blastocyst will be analyzed from each arm.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing 2nd cycle of IVF

Exclusion Criteria:

* Polycystic ovarian syndrome patient

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patient who had failed their first IVF treatment
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-03-13 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
total cumulative dosage of Gonadotropins | for 1 year duration
  number of total dosage that utilize during one cycle of IVF treatment
Total number of matured oocytes | for 1 year duration
  number of matured oocytes following the stimulation protocol
total number of good quality blastocyst | for 1 year duration
  total blastocyst achieved after each sti,ulation protocol

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Azrai Abu, MD, Principal Investigator — Department Of Obstetrics And Gynecology, Ukm Medical Centre
Locations (1):
- Advanced Reproductive Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Leahy BD, Racowsky C, Needleman D. Inferring simple but precise quantitative models of human oocyte and early embryo development. J R Soc Interface. 2021 Sep;18(182):20210475. doi: 10.1098/rsif.2021.0475. Epub 2021 Sep 8. PMID 34493094
- [Result] Simopoulou M, Sfakianoudis K, Antoniou N, Maziotis E, Rapani A, Bakas P, Anifandis G, Kalampokas T, Bolaris S, Pantou A, Pantos K, Koutsilieris M. Making IVF more effective through the evolution of prediction models: is prognosis the missing piece of the puzzle? Syst Biol Reprod Med. 2018 Oct;64(5):305-323. doi: 10.1080/19396368.2018.1504347. Epub 2018 Aug 8. PMID 30088950
- [Result] Hariton E, Chi EA, Chi G, Morris JR, Braatz J, Rajpurkar P, Rosen M. A machine learning algorithm can optimize the day of trigger to improve in vitro fertilization outcomes. Fertil Steril. 2021 Nov;116(5):1227-1235. doi: 10.1016/j.fertnstert.2021.06.018. Epub 2021 Jul 10. PMID 34256948
- [Result] Fanton M, Nutting V, Rothman A, Maeder-York P, Hariton E, Barash O, Weckstein L, Sakkas D, Copperman AB, Loewke K. An interpretable machine learning model for individualized gonadotrophin starting dose selection during ovarian stimulation. Reprod Biomed Online. 2022 Dec;45(6):1152-1159. doi: 10.1016/j.rbmo.2022.07.010. Epub 2022 Jul 28. PMID 36096871
- [Result] Correa N, Cerquides J, Arcos JL, Vassena R. Supporting first FSH dosage for ovarian stimulation with machine learning. Reprod Biomed Online. 2022 Nov;45(5):1039-1045. doi: 10.1016/j.rbmo.2022.06.010. Epub 2022 Jun 18. PMID 35915001
- [Result] Curchoe CL, Flores-Saiffe Farias A, Mendizabal-Ruiz G, Chavez-Badiola A. Evaluating predictive models in reproductive medicine. Fertil Steril. 2020 Nov;114(5):921-926. doi: 10.1016/j.fertnstert.2020.09.159. PMID 33160514